CLINICAL TRIAL: NCT03810534
Title: Connect-Home: Testing the Efficacy of Transitional Care of Patients and Caregivers During Transitions From Skilled Nursing Facilities to Home
Brief Title: Connect-Home Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-1513; R01NR017636 (NIH)
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Results first posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2021-12

CONDITIONS: Transitional Care; Caregivers; Patient Discharge; Aging; Frailty
Keywords: Transitional Care; Skilled Nursing Facilities
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: The Connect-Home study employs a stepped wedge cluster-randomized trial design, which is a crossover design at the cluster level where clusters of individuals (i.e., residents in a nursing home) crossover from control to intervention condition at randomly assigned timepoints or steps.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect-Home (Experimental): Connect-Home intervention at the skilled nursing facility and at the subject's home.
  Interventions: Behavioral: Connect-Home
- Control (No Intervention): Standard discharge planning at the skilled nursing facility only.

INTERVENTIONS:
Behavioral: Connect-Home — Connect-Home will introduce organizational structure to support delivery of transitional care processes. New elements of structure include:electronic health record (EHR) template, Connect-Home Toolkit, and Staff Training. After structural elements are added, SNF staff will use Connect-Home care processes to deliver the 2-step transitional care intervention.In Step 1, SNF nurses, therapists, and social workers will develop a Transition Plan of Care and prepare the patient and caregiver to manage the patient's serious illness and functional needs. In Step 2, the Connect-Home Activation RN will visit the patient's home within 24 hours of discharge; the nurse will activate the Transition Plan of Care at home. Both intervention steps focus on 6 key care needs to optimize patient and caregiver outcomes: 1) home safety and level of assistance; 2) advance care planning; 3) symptom management; 4) medication reconciliation; 5) function and activity; and 6) coordination of follow-up medical care.
  Arms: Connect-Home

SUMMARY:
This study will test whether transitional care targeting care needs of seriously ill, skilled nursing facility (SNF) patients and their caregivers will help to improve SNF patient outcomes (preparedness for discharge, quality of life, function and acute care use) and caregiver outcomes (preparedness for the caregiving role. caregiver burden and caregiver distress).

DETAILED DESCRIPTION:
Prior research has not established an evidence-based model of transitional care for seriously ill SNF patients (and their caregivers) who transfer from SNF to home-based care. Connect-Home, the intervention to be tested in this study, will use existing nursing home staff and community-based nurses to deliver transitional care in SNFs and the patient's home.

The feasibility, acceptability, and estimated efficacy of Connect-Home was demonstrated in a pilot test of pre-discharge elements of Connect-Home (N=133 patients and their caregivers). Compared to controls, intervention participants were significantly more prepared for discharge (higher scores on Care Transitions Measure-15) and they more frequently received individualized plans for continuing care at home. Virtually all SNF staff participants (97%) recommended the intervention for future use, demonstrating its acceptability. The objective of this study is to test the efficacy of Connect-Home for seriously ill patients discharged to home and their caregivers.

In this trial, intervention participants will receive the Connect-Home intervention; the intervention has two steps. While the patient is in the SNF, nurses, social workers and rehabilitation therapists will create an individualized Transition Plan of Care and prepare the patient and caregiver to manage the patient's serious illness at home. Within 24 hours of the time that the SNF patient discharges to home, a Connect-Home Activation Nurse (Activation RN) will visit the patient at home; the Activation RN will help the patient and family caregiver implement the written Transition Plan of Care. The Connect-Home intervention will focus on six key care needs: (1) home safety and level of assistance; (2) advance care planning; (3) symptom management; (4) medication reconciliation; (5) function and activity; and (6) coordination of follow-up medical care. In this trial, the control participants will receive usual discharge planning in the SNF only. Usual discharge planning for SNF patients includes assignment to an interdisciplinary team that develops discharge instructions for the patient to follow at home with oversight by a physician. Usual care does not include a structured home visit after the patient discharges to home.

Patient and caregiver outcomes will assessed in 7, 30, and 60 days after the patient discharged from the SNF to home. Outcomes assessors will be blinded to study group.

ELIGIBILITY:
Inclusion Criteria for patients:

* English-speaking
* Have a Minimum Data Set 3.0 Section GG Mobility Assessment Score of 3 or less, indicating the patient requires at least 25-50% assistance for functional mobility
* Be diagnosed with at least 1 serious medical illness (neurodegenerative dementia, cancer, chronic kidney disease, cirrhosis, congestive heart failure, chronic obstructive or interstitial lung disease, acute infection with sepsis, acute major motor stroke, acute coronary syndrome, acute hip fracture, diabetes with end organ complications, or intensive care for >3 days while hospitalized)
* Having a caregiver who can be enrolled in the study
* For patients with cognitive impairment additional criteria include documentation in the medical record of a caregiver who is the patient's legally authorized representative; and consent of the caregiver to participate in the study as the patient's representative.

Inclusion Criteria for Caregivers:

* English-speaking
* Self-reports assisting the patient at home.

Exclusion Criteria for Patients:

* Planned hospital readmission for procedures/treatments in next 90 days.

There are no exclusion criteria for Caregivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Toles, PhD, RN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication.
Access Criteria: Investigators who propose to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and must execute a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Toles M, Colon-Emeric C, Hanson LC, Naylor M, Weinberger M, Covington J, Preisser JS. Transitional care from skilled nursing facilities to home: study protocol for a stepped wedge cluster randomized trial. Trials. 2021 Feb 5;22(1):120. doi: 10.1186/s13063-021-05068-0. PMID 33546737

RESULTS

PARTICIPANT FLOW:
Groups:
- SNF 1: Connect-Home intervention at skilled nursing facility (SNF) 1.
  Participants at this SNF enter the Standard of Care phase for 5 months, the Pre-Implementation phase for 2 months and the Connect-Home phase for 11 months.
  Participants will encounter discharge planning at the skilled nursing facility and will have data collected at 7, 30, and 60 days post SNF discharge.
- SNF 2: Connect-Home intervention at skilled nursing facility (SNF) 2.
  Participants at this SNF enter the Standard of Care phase for 6 months, the Pre-Implementation phase for 2 months and the Connect-Home phase for 10 months.
  Participants will encounter discharge planning at the skilled nursing facility and will have data collected at 7, 30, and 60 days post SNF discharge.
- SNF 3: Connect-Home intervention at skilled nursing facility (SNF) 3.
  Participants at this SNF enter the Standard of Care phase for 7 months, the Pre-Implementation phase for 2 months and the Connect-Home phase for 9 months.
  Participants will encounter discharge planning at the skilled nursing facility and will have data collected at 7, 30, and 60 days post SNF discharge.
- SNF 4: Connect-Home intervention at skilled nursing facility (SNF) 4.
  Participants at this SNF enter the Standard of Care phase for 8 months, the Pre-Implementation phase for 2 months and the Connect-Home phase for 8 months.
  Participants will encounter discharge planning at the skilled nursing facility and will have data collected at 7, 30, and 60 days post SNF discharge.
- SNF 5: Connect-Home intervention at skilled nursing facility (SNF) 5.
  Participants at this SNF enter the Standard of Care phase for 9 months, the Pre-Implementation phase for 2 months and the Connect-Home phase for 7 months.
  Participants will encounter discharge planning at the skilled nursing facility and will have data collected at 7, 30, and 60 days post SNF discharge.
- SNF 6: Connect-Home intervention at skilled nursing facility (SNF) 6.
  Participants at this SNF enter the Standard of Care phase for 10 months, the Pre-Implementation phase for 2 months and the Connect-Home phase for 6 months.
  Participants will encounter discharge planning at the skilled nursing facility and will have data collected at 7, 30, and 60 days post SNF discharge.
Period: Standard of Care (5-10 Months)
Arm/Group | SNF 1 | SNF 2 | SNF 3 | SNF 4 | SNF 5 | SNF 6
Started | 40 | 46 | 54 | 62 | 34 | 88
Patients Started | 20 | 23 | 27 | 31 | 17 | 44
Caregivers Started | 20 | 23 | 27 | 31 | 17 | 44
Completed 7-day (Patients) | 16 | 20 | 23 | 29 | 13 | 40
Completed 7-Day (Caregivers) | 18 | 21 | 23 | 29 | 13 | 38
Completed 30-day (Patients) | 14 | 16 | 21 | 23 | 12 | 38
Completed 30-Day (Caregivers) | 14 | 16 | 21 | 23 | 10 | 32
Completed 60-Day (Patients) | 10 | 16 | 17 | 20 | 10 | 32
Completed 60-Day (Caregivers) | 10 | 16 | 15 | 20 | 9 | 31
Completed | 20 | 32 | 32 | 40 | 19 | 63
Not Completed | 20 | 14 | 22 | 22 | 15 | 25
Period: Pre-Implementation Phase (2 Months)
Arm/Group | SNF 1 | SNF 2 | SNF 3 | SNF 4 | SNF 5 | SNF 6
Started | 0 | 0 | 0 | 0 | 0 | 0
Patients Started | 0 | 0 | 0 | 0 | 0 | 0
Caregivers Started | 0 | 0 | 0 | 0 | 0 | 0
Completed 7-Day (Patients) | 0 | 0 | 0 | 0 | 0 | 0
Completed 7-Day (Caregivers) | 0 | 0 | 0 | 0 | 0 | 0
Completed 30-Day (Patients) | 0 | 0 | 0 | 0 | 0 | 0
Completed 30-Day (Caregivers) | 0 | 0 | 0 | 0 | 0 | 0
Completed 60-Day (Patients) | 0 | 0 | 0 | 0 | 0 | 0
Completed 60-Day (Caregivers) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Connect-Home (5-10 Months)
Arm/Group | SNF 1 | SNF 2 | SNF 3 | SNF 4 | SNF 5 | SNF 6
Started | 82 | 80 | 66 | 54 | 10 | 38
Patients Started | 41 | 40 | 33 | 27 | 5 | 19
Caregivers Started | 41 | 40 | 33 | 27 | 5 | 19
Completed 7-Day (Patients) | 38 | 35 | 27 | 23 | 4 | 14
Completed 7-Day (Caregivers) | 35 | 34 | 29 | 24 | 4 | 13
Completed 30-Day (Patients) | 35 | 31 | 25 | 19 | 3 | 12
Completed 30-Day (Caregivers) | 34 | 30 | 25 | 21 | 2 | 10
Completed 60-Day (Patients) | 30 | 25 | 23 | 19 | 2 | 10
Completed 60-Day (Caregivers) | 32 | 27 | 21 | 19 | 2 | 9
Completed | 62 | 52 | 44 | 38 | 4 | 19
Not Completed | 20 | 28 | 22 | 16 | 6 | 19

BASELINE CHARACTERISTICS:
Groups:
- Connect-Home Patients: Connect-Home intervention at the skilled nursing facility and at the subject's home. Participants will have data collected at 7, 30, and 60 days post SNF discharge.
- Connect-Home Caregivers: Caregivers of Connect-Home study patients.
- Control Patients: Standard discharge planning at the skilled nursing facility only. Participants will have data collected at 7, 30, and 60 days post SNF discharge.
- Control Caregivers: Caregivers of Control study patients.
- Total: Total of all reporting groups
Arm/Group | Connect-Home Patients | Connect-Home Caregivers | Control Patients | Control Caregivers | Total
Number analyzed (Participants) | 165 | 165 | 162 | 162 | 654
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.5 (9.49) | 58.1 (14.02) | 76.6 (9.55) | 60.9 (13.72) | 76.5 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 119 | 105 | 116 | 444
  Male | 61 | 46 | 57 | 46 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 165 | 165 | 162 | 162 | 654
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 37 | 37 | 40 | 43 | 157
  White | 123 | 117 | 119 | 113 | 472
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 11 | 3 | 6 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 165 | 165 | 162 | 162 | 654

OUTCOME MEASURES:

1. Primary Outcome: Care Transitions Measure-15 Score 7 Days After Skilled Nursing Facility Discharge
Description: The patient's preparedness for discharge will be measured by the Care Transitions Measure-15 (CTM-15), which includes 5 items on a 4-point scale. The CTM-15 measures self-reported knowledge and skills for continuing care at home. Summary score range 0-100, with higher scores associated with less acute care use after discharge.
Time Frame: 7 Days After SNF Discharge
Population: Data reported for participants who answered the 7-day data collection phone call.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Connect-Home: Connect-Home intervention at the skilled nursing facility and at the subject's home. Participants will have data collected at 7, 30, and 60 days post SNF discharge.
- Control: Standard discharge planning at the skilled nursing facility only. Participants will have data collected at 7, 30, and 60 days post SNF discharge
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 142 | 141
score on a scale | 75.80 (16.08) | 68.33 (17.69)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .62, Mixed Models Analysis; Mean Difference (Final Values) = -1.64, Standard Error of Mean 3.24 — The final estimated mean difference is based on a linear mixed model that adjusts for time and is not equal to the difference in the unadjusted, observed means

2. Primary Outcome: Preparedness for Caregiving Scale Score 7 Days After Patient's Skill Nursing Facility Discharge
Description: The caregiver's preparedness for caregiving will be measured by the Preparedness for Caregiving Scale (PCS), which includes 8 items on a five-point Likert scale (0-4). The PCS measures self-reported readiness for caregiving. Range = 0-32, with higher scores associated with less anxiety.
Time Frame: 7 Days After Patient SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 140 | 141
score on a scale | 23.14 (6.74) | 19.26 (6.42)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .31, Mixed Models Analysis; Mean Difference (Final Values) = -1.47, Standard Error of Mean 1.44 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: McGill Quality of Life Questionnaire-Revised Score 30 Days After Skilled Nursing Facility Discharge
Description: The patient's quality of life will be measured using the McGill Quality of Life Questionnaire-Revised (MQoL-R), which includes 14 items on a ten-point Likert scale. The scale is recommended for studies of palliative care and measures quality of life across disease trajectories. Range = 0-10, with higher score indicating better quality of life. There are 4 MQOL-R subscales. Each subscale score is the mean of its items that range from 0-10. The Total Score, also ranging from 0-10, is the mean of the subscale score means.
Time Frame: 30 Days After SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 100 | 91
score on a scale | 7.69 (1.81) | 7.69 (1.79)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .93, Mixed Models Analysis; Mean Difference (Final Values) = .03, Standard Error of Mean .33 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: McGill Quality of Life Questionnaire-Revised Score 60 Days After Skilled Nursing Facility Discharge
Description: as for outcome 3
Time Frame: 60 Days After SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 88 | 81
score on a scale | 7.81 (1.58) | 7.71 (1.73)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .60, Mixed Models Analysis; Mean Difference (Final Values) = .18, Standard Error of Mean .34 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Life Space Assessment 30 Days After Skilled Nursing Facility Discharge
Description: Patient's function will be measured using the Life Space Assessment, which includes 5 Likert scales corresponding to a hierarchy of levels of mobility (each scored from 0-4) where weights are the product of the "Life-space level" (range 1-5) and the "independence" score (range 1-2). The range is 1-120. Lower scores are associated with falls and hospitalization.
Time Frame: 30 Days After SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 124 | 125
score on a scale | 22.18 (16.67) | 22.97 (15.38)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .53, Mixed Models Analysis; Mean Difference (Final Values) = 2.24, Standard Error of Mean 3.49 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Life Space Assessment 60 Days After Skilled Nursing Facility Discharge
Description: as for outcome 5
Time Frame: 60 Days After SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 108 | 105
score on a scale | 25.55 (17.41) | 28.60 (18.55)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .83, Mixed Models Analysis; Mean Difference (Final Values) = .78, Standard Error of Mean 3.57 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Zarit Caregiver Burden Scale 30 Days After Skilled Nursing Facility Discharge
Description: Caregiver burden will be measured using the Zarit Caregiver Burden Scale, which includes 12 items on a five-point scale, measuring caregiver perceptions that "caregiving has an adverse effect on their emotional, social, financial, physical and spiritual functioning." Scores range 0-48; higher scores are associated with depression and social isolation.
Time Frame: 30 Days After Patient's SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 120 | 118
score on a scale | 12.27 (9.77) | 12.33 (10.33)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .75, Mixed Models Analysis; Mean Difference (Final Values) = .67, Standard Error of Mean 2.05 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Zarit Caregiver Burden Scale 60 Days After Skilled Nursing Facility Discharge
Description: as for outcome 7
Time Frame: 60 Days After Patient's SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 106 | 102
score on a scale | 11.84 (9.40) | 11.35 (8.94)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .50, Mixed Models Analysis; Mean Difference (Final Values) = 1.44, Standard Error of Mean 2.07 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Distress Thermometer 30 Days After Skilled Nursing Facility Discharge
Description: Caregiver distress will be measured using the Distress Thermometer, which includes 1 item on an 11-point scale, measuring negative affect (e.g., sadness and fear) related to caregiving for a severely ill person. Score ranges 0-10, with scores >4 associated with poor coping and depression.
Time Frame: 30 Days After Patient's SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 118 | 118
score on a scale | 3.19 (2.66) | 3.02 (3.08)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .48, Mixed Models Analysis; Mean Difference (Final Values) = .36, Standard Error of Mean .50 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Distress Thermometer 60 Days After Skilled Nursing Facility Discharge
Description: as for outcome 9
Time Frame: 60 Days After Patient's SNF Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 105 | 102
score on a scale | 3.03 (3.07) | 2.60 (2.73)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .22, Mixed Models Analysis; Mean Difference (Final Values) = .65, Standard Error of Mean .52 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Self-Reported Days of ED or Hospital Use 30 Days After Skilled Nursing Facility Discharge
Description: Patient's days of acute care use will be measured using the self-reported number of combined number of days the patient spends in the Emergency Department (ED) or hospital in 30 days after SNF discharge.
Time Frame: 30 Days After SNF Discharge
Population: Data are reported only for participants who had acute care use.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 135 | 130
Days | .65 (1.82) | 1.01 (3.46)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .88, Mixed Models Analysis; Mean ratio = .96, Standard Error of Mean .25

12. Secondary Outcome: Self-Reported Days of ED or Hospital Use 60 Days After Skilled Nursing Facility Discharge
Description: Patient's days of acute care use will be measured using the self-reported number of combined number of days the patient spends in the ED or hospital in 60 days after SNF discharge.
Time Frame: 60 Days After SNF Discharge
Population: Data are reported only for participants who had acute care use.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Connect-Home | Control
Number analyzed (Participants) | 136 | 131
Days | .82 (2.00) | 1.24 (3.61)
Statistical Analysis 1: Comparison: Connect-Home vs Control; Test type: Superiority; p = .23, Mixed Models Analysis; Mean ratio = .72, Standard Error of Mean .18

ADVERSE EVENTS:
Time Frame: Adverse events were collected from when participants entered the study to when they completed study procedures, an approximate total of up to 90 days.
Description: Due to the severity of illness present in the study population, unrelated adverse events were expected during this study.
Arm/Group | Connect-Home Patients | Connect-Home Caregivers | Control Patients | Control Caregivers
All-Cause Mortality (participants affected / at risk) | 6/165 | 0/165 | 8/162 | 0/162
Serious Adverse Events (participants affected / at risk) | 38/165 | 0/165 | 34/162 | 0/162
Other Adverse Events (participants affected / at risk) | 0/165 | 0/165 | 0/162 | 0/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Connect-Home Patients (N=165) | Connect-Home Caregivers (N=165) | Control Patients (N=162) | Control Caregivers (N=162)
Hospitalization for generalized weakness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Reason Undisclosed (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Hospitalization for Racing Heart Issues (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization for Neck Laceration Caused by Fall (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization due to Mini Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hospitalization due to Urinary Tract Infection (Renal and urinary disorders) | 5 (5) | 0 (0) | 4 (4) | 0 (0)
Hospitalization due to Kidney Issues (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Acute Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Hospitalization Due to Low Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Fluid Build-Up (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Left Thoracentesis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Fracture Subsequent to Fall (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0) | 4 (4) | 0 (0)
Hospitalization Due to Gall Bladder Issues (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Cardiac Stent Placement (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Skin Infection (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Colon Tear (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalization Due to Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Hospitalization Due to Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Pulmonary Embolism (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Lower Extremity Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Tremors (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Toe Amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hospitalization Due to Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization Due to Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03810534/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT03810534/ICF_001.pdf